CLINICAL TRIAL: NCT03025191
Title: Development and Acceptability Evaluation of a Novel STI/HIV Prevention Intervention for Couples Affected by Incarceration
Brief Title: Prison Connect-STI/HIV Prevention Intervention for Couples Affected by Incarceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Yale University (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-00604
Record Dates: First submitted 2017-01-17; First posted 2017-01-19 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2017-12

CONDITIONS: Incarceration
Keywords: incarceration; HIV
MeSH Terms: interventions — Organizational Objectives

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prison Connect (Experimental)
  Interventions: Behavioral: Speaker/Listener technique; Behavioral: Social Support; Behavioral: Problem-Solving; Behavioral: Goal Setting

INTERVENTIONS:
Behavioral: Speaker/Listener technique — Couple will learn taking turns as the speaker and as the listener who paraphrases the speaker's point.The couple will then identify an issue they have faced in their relationship and will role-play using the technique to discuss it.
Behavioral: Social Support — Identification of and mapping sources of social support and the types of support provided by members of the network. Participants will also identify the strengths and weaknesses of their support network and think through ways to strengthen those networks.
Behavioral: Problem-Solving — Couple will be taught steps to systematically analyze a problem and brainstorm solutions through a short video. Steps include identify the trigger/problem; identify the goal for addressing the problem; brainstorm possible solutions for each partner; evaluate the solutions and pick the best; and act on the best solution.
Behavioral: Goal Setting — Couple will be introduced to the concept of short- and long-term goal setting, including components of goal and planning for potential barriers. The couple will then set a goal for themselves that incorporates the skills obtained during the intervention, such as strengthening ties in their social support network. Participants will fill in a worksheet outlining their goal, potential barriers, and solutions to those barriers.

SUMMARY:
The purpose of this study is to adapt an existing couples-level HIV prevention intervention for community populations (CONNECT I/II; PI: El-Bassel) to enable implementation among couples affected by incarceration (PRISON CONNECT) and pilot test its feasibility and acceptability among men incarcerated in the Connecticut Department of Correction (CTDOC) and their community-dwelling committed female partners.

DETAILED DESCRIPTION:
This pilot study will recruit male inmates in the Connecticut Department of Correction and their community-dwelling female partner. Using an adapted version of an efficacious couples-level HIV prevention intervention for community populations (CONNECT; PI: El-Bassel), this study will pilot test a single in-prison intervention session using face-to-face or teleconferencing modalities and a brief community follow-up session. Feasibility and acceptability among the inmates and their partners will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* eight HIV-positive and HIV-negative/unknown status male inmates and their partners (N=16 couples, 32 participants).

Male Participants

* at least 18 years of age
* able to communicate in English, currently
* incarcerated in the Connecticut Department of Correction (CTDOC), due to be released within three months.
* have a committed female partner who is not currently incarcerated and willing to participate in the study, and is
* not concerned participation will cause violence in the relationship.

Female partners

* be able to communicate in English
* not currently incarcerated
* confirm the committed partnership with the male inmate and willingness to participate in the study
* not concerned participation in the study would cause violence in the relationship.

Exclusion Criteria:

* restricted to English-speaking participants due to language availability of staff and intervention materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Acceptability of intervention procedures and content by administration of a brief acceptability questionnaire among incarcerated men and their partners | 15 Minutes
  Questions about how participant feels about the program activities.

SECONDARY OUTCOMES:
Acceptability of follow-up procedures and follow-up intervention content by administration of a brief acceptability questionnaire among male releasees and their partners. | 15 Minutes
  Using tracking information provided at the time of in-prison session of PRISON CONNECT investigators will initiate contact with couples within the first month of release and conduct the follow-up visit at a location/time convenient for couples (e.g., team's research facility in New Haven, CT). The session will include a review of PRISON CONNECT intervention content.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Khan, MD, Principal Investigator — New York University Medical School
Locations (1):
- New York University School of Medicine, New York, New York, United States